CLINICAL TRIAL: NCT04043195
Title: Nivolumab (Anti-PD1 Antibody) and Ipilimumab (Anti-CTLA4 Antibody) in Combination With Immunogenic Chemotherapy for Patients With Advanced Non-Small Cell Lung Cancer
Brief Title: Nivolumab and Ipilimumab in Combination With Immunogenic Chemotherapy for Patients With Advanced NSCLC
Acronym: NSCLC
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hatim Husain (Other)
Responsible Party: Sponsor-Investigator, Hatim Husain, Associate Professor, University of California, San Diego
Organization: University of California, San Diego (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 181485
Record Dates: First submitted 2019-07-25; First posted 2019-08-02 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Advanced NSCLC
Keywords: NSCLC; Ipilimumab; Nivolumab; Oxaliplatin
MeSH Terms: interventions — Nivolumab; Oxaliplatin; Ipilimumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Nivolumab + Oxaliplatin + Ipilimumab (Experimental): Cohort 1
  Interventions: Drug: Nivolumab; Drug: Oxaliplatin; Drug: Ipilimumab

INTERVENTIONS:
Drug: Nivolumab — 240 mg every 2 weeks. Nivolumab will continue for up to 2 years.
  Other Names: Opdivo
Drug: Oxaliplatin — 65 mg/m2 every 2 weeks. Oxaliplatin will continue for up to 12 cycles.
  Other Names: Eloxatin
Drug: Ipilimumab — 1 mg/kg every 6 weeks. Ipilimumab will continue for up to 4 cycles
  Other Names: Yervoy

SUMMARY:
The purpose of this study is to examine the safety and efficacy of combining Nivolumab and low-dose Oxaliplatin with or without Ipilumumab in patients who have had their advanced NSCLC cancer worsen on or after being treated with certain immunotherapies (drugs that target the immune system).

DETAILED DESCRIPTION:
The purpose of this study is to examine the safety and efficacy of combining Nivolumab and low-dose Oxaliplatin with or without Ipilumumab in patients who have had their advanced NSCLC cancer worsen on or after being treated with certain immunotherapies (drugs that target the immune system).

Nivolumab (Opdivo®) is approved by the Food and Drug Administration (FDA) for the treatment of metastatic (the cancer has spread) NSCLC. It is a type of drug called a monoclonal antibody (a type of protein). Monoclonal antibodies bind to other proteins, such as PD-1 (programmed cell death-1), on immune cells, which allows the immune cells to continue working against the tumor.

Ipilumumab (Yervoy®) is also a monoclonal antibody, but binds to a protein called CTLA-4 (cytotoxic T-lymphocyte-associated protein 4).

Oxaliplatin is a type of immunogenic chemotherapy, which may increase the body's immune response to the cancer. Both are approved for treatment of other types of cancers, but not in patients with NSCLC.

ELIGIBILITY:
The following list is a summary. Additional criteria apply.

Inclusion Criteria:

Patients must meet all of the following criteria to be eligible for study entry.

* At least 18 years or older
* Histologically or cytologically confirmed, advanced non-squamous or squamous NSCLC
* Last line of therapy for advanced non-squamous or squamous NSCLC must be with an anti-PD1 or PDL1 antibody with confirmed progression on or after that treatment. Patients may have received no more than 3 lines of prior therapy including no more than 2 prior lines of therapy containing a PD-(L)-2 antibody. Patients must have received prior cisplatin or carboplatin based doublet chemotherapy.
* Measurable disease, as defined by RECIST v1.1
* Adequate hematologic and end-organ function, defined by the laboratory test results within 14 days prior to randomization:
* For female patients of childbearing potential and male patients with partners of childbearing potential, agreement to use a highly effective form(s) of contraception during study treatment that results in a low failure rate of <1% per year when used consistently and correctly. Female patients should continue contraception use for 5 months after the last dose of nivolumab and ipilimumab and for 6 months after the last dose of oxaliplatin. Make patients treated with chemotherapy should continue contraception use for 7 months after the last dose of chemotherapy. Men should refrain from donating sperm during this same period. Such methods include combined (estrogen and progestogen containing) hormonal contraception, with another additional barrier method always containing a spermicide, intrauterine device (IUD), intrauterine hormone-releasing system (IUS), bilateral tubal occlusion or vasectomized partner (on the understanding that this is the only one partner during the study duration), and sexual abstinence.

  * Oral contraception should always be combined with an additional contraceptive method because of a potential interaction with the study drug. The same rules are valid for male patients involved in this study if they have a partner of childbearing potential. Male patients must always use a condom.
  * Women who are not postmenopausal (>12 months of non-therapy-induced amenorrhea) or surgically sterile must have a negative serum pregnancy test result within 14 days prior to initiation of study drug.

Exclusion Criteria:

General Medical Exclusions

* Women who are pregnant, lactating, or intending to become pregnant during the study.
* History of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric or humanized antibodies or fusion proteins.
* History of autoimmune disease
* History of idiopathic pulmonary fibrosis, organizing pneumonia (e.g. bronchiolitis obliterans), drug-induced pneumonitis, idiopathic pneumonitis, or evidence of active pneumonitis on screening chest CT scan.
* Major surgical procedure other than for diagnosis within 28 days prior to randomization or anticipation of need for a major surgical procedure during the course of the study.
* Prior allogeneic bone marrow transplantation or solid organ transplantation.

Exclusion Criteria Related to Medications

* Treatment with any approved anti-cancer therapy within 2 weeks prior to initiation of study treatment.
* Treatment with any other investigational agent with therapeutic intent within 21 days prior to enrollment.
* Received therapeutic oral or intravenous (IV) antibiotics within 2 weeks prior to enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-08-14 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | 4 months
  To estimate ORR by RECIST 1.1

SECONDARY OUTCOMES:
Overall survival (OS) | 1 and 2 year
  Overall survival (OS)
Progression-free survival (PFS) | 1 year
  Progression-free survival (PFS)

CONTACTS AND LOCATIONS:
Overall Officials: Hatim Husain, Principal Investigator — University of California, San Diego
Locations (1):
- UC San Diego Moores Cancer Center, La Jolla, California, United States